CLINICAL TRIAL: NCT03581019
Title: Uterus Transplantation From Deceased Donor - Gothenburg III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Brännström, Professor, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sahlgrenska-DD-UTx
Record Dates: First submitted 2018-06-17; First posted 2018-07-10 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Absolute Uterine Factor Infertility; Transplantation; Mrk Anomaly
Keywords: infertility, uterus, transplantation, MRKH
MeSH Terms: conditions — Mullerian aplasia; Infertility

STUDY DESIGN:
Intervention Model Description: Observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterus transplantation (Experimental): Uterus transplantation
  Interventions: Procedure: uterus transplantation

INTERVENTIONS:
Procedure: uterus transplantation — uterus transplantation from deceased donor

SUMMARY:
Deceased donor uterus transplantation will be offered to patients that have either been excluded from Gothenburg II because of donor criteria or because of early graft failure in Gothenburg I and II

ELIGIBILITY:
Inclusion criteria recipient

* initially included with IVF and excluded by donor issues of Gothenburg I or II
* initially included and excluded by early graft failure of Gothenburg I or II
* age < 40 years
* no systemic disease
* no standing medication
* satisfactory ovarian reserve
* BMI <35 and at BMI 30-35 waist circumference of < 82 cm
* absolute uterine factor infertility
* psychological stable

Inclusion criteria donor

* brain death and suitable as multiorgan donor
* acceptance for donation of uterus from family or previously by patient
* age <55 years
* at least one normal pregnancy and childbirth
* no previos malignancy
* no systemic disease
* no previous major surgery inn abdomen or on uterus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
birth of healthy child | 1-5 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mats Brännström, Principal Investigator — Göteborg University
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Mats Brännström, Gothenburg